CLINICAL TRIAL: NCT02613481
Title: The Emotional and Functional Benefits of Poly-L-Lactic Acid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yardley Dermatology Associates (Other)
Collaborators: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: YDA-001
Record Dates: First submitted 2015-10-29; First posted 2015-11-24 (Estimated); Results first posted 2019-05-29 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Facial Volume Loss
MeSH Terms: interventions — poly(lactide); New-Fill; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Poly-L-Lactic Acid (Sculptra) injection (Other): Poly-L-Lactic Acid (Sculptra) injection for all enrolled subjects
  Interventions: Drug: Poly-L-Lactic Acid (Sculptra) injection

INTERVENTIONS:
Drug: Poly-L-Lactic Acid (Sculptra) injection — 1 vial of of poly-l-lactic acid (Sculptra) reconstituted in the usual sterile fashion with 7cc of sterile water and 2cc of Lidocaine without epinephrine. The contents of the vial will be injected as deemed appropriate by the certified injector and agreed upon by the study subject.

SUMMARY:
This study will evaluates the emotional and functional benefits of Poly-L-Lactic Acid (Sculptra™), a cosmetic product used to fill defects of the skin. All participants will receive Sculptra™.

DETAILED DESCRIPTION:
Facial volume loss can result in emotional distress and functional impairment in some affected individuals. Poly-L-Lactic Acid (Sculptra™) stimulates collagen production in the skin thereby replenishing some of the collagen lost to natural aging and ultraviolet damage. This study will assess the emotional and functional benefits of Poly-L-Lactic Acid treated subject's through self report measurement tools.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be an outpatient, male or female subjects of any race, 35 years of age or older.
2. Subject must have any degree of facial volume loss.
3. Subjects of all Fitzpatrick skin types are eligible.
4. Subject must be able to follow study instructions and likely to complete all required visits, as assessed by the Investigator.
5. Subject must sign an IRB-approved Informed Consent form, Photographic Release Form, and the Authorization for Use and release of Health and Research Study Information (HIPAA) form prior to any study-related procedures being performed.

Exclusion Criteria:

1. Any of the previous facial treatments:

   c. Any facial filler in the past 2 years d. Prior injection of permanent facial implant
2. Have any skin pathology or condition that could interfere with the evaluation of the face.
3. Be unable to communicate or cooperate with the Investigator due to a language barrier (non-English speaking), poor mental development, or impaired cerebral function.
4. Have evidence of alcohol or drug abuse (Investigator opinion), or history of poor cooperation, non-compliance with medical treatment, or unreliability.
5. Have used an investigational device, biologic or drug in the past 30 days, or be currently participating in an experimental drug, biologic or device trial.
6. Have a condition or be in a situation that, in the Investigator's opinion, may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study.
7. Be an employee (or a relative of an employee) of the Investigator, Sponsor or representative of the Sponsor.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-11; Primary Completion 2017-06-01 (Actual); Study Completion 2017-08-01 (Actual)

REFERENCES:
- See also: Click here for more information about this study: The Emotional and Functional Benefits of Poly-L-Lactic Acid — http://yardleyderm.com//

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Poly-L-Lactic Acid (Sculptra) Injection
Started | 50
Completed | 41
Not Completed | 9
Not completed — Lost to Follow-up | 7
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Poly-L-Lactic Acid (Sculptra) Injection
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 43
  >=65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49
  Male | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 2
  Ethnicity: Non Hispanic or Latino | 47
  Ethnicity: American Indian or Alaskan | 1
  Ethnicity: Hawaiian or Pacific Islander | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Mean Subject Self Reported Quality of Life Scale
Description: Self report Likert Scale Title: Facial Volume Restoration Outcome Questionnaire 35 Questions 1-7 rating with higher score meaning a worse outcome
Time Frame: 3 months post initial injection
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Poly-L-Lactic Acid (Sculptra) Injection
Number analyzed (Participants) | 50
units on a scale | 3.45 (0.39)

2. Primary Outcome: Mean Rosenberg Self-Esteem Scale
Description: Self reported self esteem measure Title: Rosenberg Self-Esteem Scale Scale of 1-4, scale design with higher score relating to worse outcome.
Time Frame: 3 months post initial injection
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Poly-L-Lactic Acid (Sculptra) Injection
Number analyzed (Participants) | 50
units on a scale | 2.56 (.93)

3. Primary Outcome: Mean Rosenberg Self-Esteem Scale
Description: as for outcome 2
Time Frame: 6 months post initial injection
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Poly-L-Lactic Acid (Sculptra) Injection
Number analyzed (Participants) | 50
units on a scale | 2.24 (1.05)

4. Primary Outcome: Mean Subject Self Reported Quality of Life Scale
Description: as for outcome 1
Time Frame: 6 months post initial injection
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Poly-L-Lactic Acid (Sculptra) Injection
Number analyzed (Participants) | 50
units on a scale | 3.22 (0.37)

ADVERSE EVENTS:
Time Frame: 9 Months
Description: Subject population of decreased facial volume not due to concomitant disease state is not considered at higher risk for mortality than age matched general population. In additional Poly-L -Lactic Acid has not been associated with any increased risk of mortality.
Arm/Group | Poly-L-Lactic Acid (Sculptra) Injection
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 5/50
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Poly-L-Lactic Acid (Sculptra) Injection (N=50)
Pain/Discomfort (Skin and subcutaneous tissue disorders) | 5 (5) — expected post procedure pain/discomfort

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-10-21): https://cdn.clinicaltrials.gov/large-docs/81/NCT02613481/Prot_SAP_000.pdf